CLINICAL TRIAL: NCT01679769
Title: Prospective Study In Noninvasive Evaluation of Hepatic Fibrosis in Chronic
Brief Title: Prospective Study In Noninvasive Evaluation of Hepatic Fibrosis in Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, Professor, Peking University First Hospital
Other Study IDs: 2012-455; 81170386 (Other Grant/Funding Number: from The National Natural Science Foundation of China)
Record Dates: First submitted 2012-09-01; First posted 2012-09-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — liver biopsy samples and blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of our study is to evaluate liver fibrosis using biochemical markers, FibroScan, and radiology methods in patients with chronic hepatitis B in mainland China.

DETAILED DESCRIPTION:
Up to Nov, 2015, total of 818 patients with chronic HBV infection had been enrolled in the study. Paired blood and liver biopsy specimen had been collected. The serum samples stored at -80 degree Celsius. All the liver biopsy samples were judged by three pathology experts, according to Ishak standard.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic hepatitis B or compensated cirrhosis due to chronic hepatitis B virus infection
* agree to have liver biopsy

Exclusion Criteria:

* clinical diagnosis of decompensated cirrhosis due to hepatitis B virus or inactive carrier
* liver diseases due to other origin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic hepatitis B or compensated cirrhosis due to chronic hepatits B virus (HBV) infection
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2012-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of staging fibrosis with a combination of non-invasive parameters compared to liver biopsy | within two weeks after liver biopsy

SECONDARY OUTCOMES:
Evaluation of staging inflammation with a combination of non-invasive parameters compared to liver biopsy | within two weeks after liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, MD, Principal Investigator — Peking University First Hospital; Hong Zhao, MD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China